CLINICAL TRIAL: NCT06931210
Title: Study of AI-based Prediction Models for Exercise-Induced Gut Microbiota Alterations in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-KY-121(K)
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Experimental)
  Interventions: Behavioral: Exercise intervention
- Sedentary control group (Other)
  Interventions: Other: Sedentary behavior

INTERVENTIONS:
Other: Sedentary behavior — Patients in the control group will maintain their sedentary lifestyle unchanged.
  Arms: Sedentary control group
Behavioral: Exercise intervention — The intervention will include a combination of aerobic and resistance exercises, performed three times per week. Each session will last 80 minutes. Aerobic and resistance training will include cycling, chest press, rowing, abdominal and back muscle exercises, as well as leg strength training.
  Arms: Exercise intervention group

SUMMARY:
This study is a randomized controlled clinical trial. The participants will be randomized into two groups in a 1:1 ratio: exercise intervention and sedentary control group. The participants (50 participants per group) will undergo a 16-week intervention. Participants in the control group will maintain their sedentary lifestyle unchanged, and the exercise intervention group will receive combined aerobic and resistance exercise training. This study aims to compare the changes in gut microbiota before and after exercise intervention in patients. It will validate and optimize a cross-species microbiota mapping model through an independent exercise intervention clinical trial. Additionally, it will comprehensively assess the effects of combined aerobic and resistance exercise on patients' body composition, the severity of fatty liver, and glucose-lipid metabolism indicators. The study will also analyze the correlation between dynamic changes in the gut microbiota and the improvement of clinical symptoms in patients with type 2 diabetes after exercise intervention, elucidating the regulatory mechanisms of microbiota remodeling in exercise-mediated metabolic benefits.

ELIGIBILITY:
Inclusion Criteria:

-1. Diagnosed with type 2 diabetes; 2. Taking ≤3 types of antidiabetic medications; 3. On a stable medication regimen for at least 6 weeks prior to the intervention and maintaining the same regimen during the study period; 4. Aged between 35 and 65 years; 5. Abdominal obesity: waist circumference >90 cm for men and >85 cm for women; 6. Body mass index (BMI) ≤35 kg/m²; 7. Waist-to-thigh ratio (WTR): ≥1.7 for men and ≥1.6 for women; 8. Sedentary lifestyle (engaging in moderate-intensity exercise for ≤60 minutes per week).

Exclusion Criteria:

-1. Glycated hemoglobin (HbA1c) <6.5% or ≥9%; 2. Use of insulin; 3. Presence of one or more of the following complications: advanced diabetic retinopathy, macroalbuminuria (urine albumin-to-creatinine ratio ≥300 mg/g), or renal dysfunction (estimated glomerular filtration rate [eGFR] ≤60 mL/min/1.73 m²); 4. History of cardiovascular events (e.g., myocardial infarction, stent implantation, unstable angina, heart failure, or cardiac dysfunction); 5. History of cerebrovascular disease (e.g., cerebral hemorrhage or ischemic stroke); 6. Muscular, skeletal, or neuromuscular injuries that hinder exercise training; 6. Severe osteoporosis or failure to meet bone mineral density criteria despite treatment; 7. Pregnancy; 8. Inability or unwillingness to undergo MRI examination (e.g., due to claustrophobia, implantable cardioverter-defibrillator [ICD], or pacemaker); 9. Diagnosed depression or any psychiatric disorder that prevents the patient from understanding the nature, scope, and possible sequence of the study; 10. Patients taking antihypertensive or lipid-lowering medications are excluded if their medication regimen is unstable or affects glucose metabolism.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota | Baseline and 16 weeks
  Gut microbiota, including microbial composition, diversity, functional metabolism, etc., will be measured at baseline and at 16 weeks using metagenomic sequencing and other related methods.

SECONDARY OUTCOMES:
Changes in body composition | Baseline and 16 weeks
  The body composition parameters, including fat mass, changes in lean mass and its percentage, abdominal and thigh fat mass, as well as hip and lower limb muscle mass, etc., will be measured at baseline and after 16 weeks.
Change in insulin sensitivity | Baseline and 16 weeks
  Insulin sensitivity will be assessed at baseline and 16 weeks.
Change in HbA1c | Baseline and 16 weeks
  HbA1c will be measured at baseline and 16 weeks. HbA1c will be expressed in mmol/mol.
Change in obesity-related anthropometrics | Baseline, 4, 8, 12, 16 weeks
  Obesity-related anthropometrics, including waist, hip, and thigh circumference, etc., will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in body mass index (BMI) | Baseline, 4, 8, 12, 16 weeks
  Height, weight and BMI will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in other indicators of glucose metabolism | Baseline, 4, 8, 12, and 16 weeks
  Other indicators of glucose metabolism, including blood glucose, insulin, C-peptide, and other relevant parameters, will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in intrahepatic triglyceride content | Baseline, 16 weeks
  Intrahepatic triglyceride content will be assessed at baseline and 16 weeks.
Change in other indicators of lipid metabolism | Baseline, 4, 8, 12, and 16 weeks
  Other indicators of lipid metabolism, including TC, TG, LDL-C, HDL-C and other relevant parameters, will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in inflammatory markers | Baseline, 4, 8, 12, and 16 weeks
  Inflammatory markers, including CRP, serum amyloid A and other relevant parameters, will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in liver function | Baseline, 4, 8, 12, and 16 weeks
  Liver function biomarkers, including ALT, AST and other relevant parameters, will be assessed at baseline, 4, 8, 12, and 16 weeks.
Change in cytokines | Baseline, 16 weeks
  Cytokines, including FGF21, FGF19, FABP4, LCN2, adiponectin, and others, will be assessed at baseline and at 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China